CLINICAL TRIAL: NCT05696847
Title: A Safety, Tolerability and Pharmacokinetic Study of Tirzepatide for the Treatment of Pediatric Participants (6 Years to 11 Years) With Obesity
Brief Title: A Study of Tirzepatide (LY3298176) in Pediatric Participants With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17370; I8F-MC-GPHV (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-01-17; First posted 2023-01-25 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Pediatrics; Obesity; Chronic weight management
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Placebo (BW >=50 kg) (Placebo Comparator): Participants in this cohort had a screening body weight (BW) of at least 50 kilograms (kg) received placebo administered subcutaneously (SC) once weekly (QW) during Weeks 1 to 8.
  Interventions: Drug: Placebo
- Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) (Experimental): Participants in this cohort had a screening body weight of at least 50 kg received 2.5 milligrams (mg) tirzepatide administered SC QW during Weeks 1 to 4 followed by 5 mg tirzepatide during Weeks 5 to 8.
  Interventions: Drug: Tirzepatide
- Cohort 2: Placebo (BW <50 kg) (Placebo Comparator): Participants in this cohort had a screening body weight less than 50 kg received placebo administered SC QW during Weeks 1 to 8.
  Interventions: Drug: Placebo
- Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) (Experimental): Participants in this cohort had a screening body weight less than 50 kg received 1.25 mg tirzepatide administered SC QW during Weeks 1 to 4 followed by 2.5 mg tirzepatide during Weeks 5 to 8.
  Interventions: Drug: Tirzepatide
- Cohort 3: Placebo (BW 40 to 60 kg) (Placebo Comparator): Participants in this cohort had a screening body weight between 40 to 60 kg, inclusive, received placebo administered SC QW during Weeks 1 to 8.
  Interventions: Drug: Placebo
- Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg) (Experimental): Participants in this cohort had a screening body weight between 40 to 60 kg, inclusive, received 2.5 mg tirzepatide administered SC QW during Weeks 1 to 4 followed by 5 mg tirzepatide during Weeks 5 to 8.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg); Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg); Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
Drug: Placebo — Administered SC
  Arms: Cohort 1: Placebo (BW >=50 kg); Cohort 2: Placebo (BW <50 kg); Cohort 3: Placebo (BW 40 to 60 kg)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of tirzepatide (LY3298176) in pediatric participants with obesity. The blood tests will be performed to investigate how the body processes the study drug in these participants. For each participant, the study will last about approximately 13 weeks excluding the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with body mass index (BMI) ≥ the 95th percentile for age and sex
* Have failed to achieve adequate weight loss through lifestyle modification in the investigator's opinion
* Female participants only: Determined as prepubertal Tanner Stage 1.

Exclusion Criteria:

* Change in body weight above 5 kg (11 lbs) within 90 days before screening irrespective of medical records
* Have obesity induced by other endocrinologic disorders (for example, Cushing syndrome) or diagnosed monogenetic or syndromic forms of obesity
* Have acute or chronic pancreatitis or a history of acute idiopathic pancreatitis; or have other GI disorders
* Have a known clinically significant gastric emptying, have undergone weight loss surgery such as gastric bypass (bariatric) surgery or restrictive bariatric surger, or have endoscopic or device-based therapy for obesity or have had device removal within the last 6 months.
* Have confirmed type 1 or type 2 diabetes mellitus
* Have a history or current cerebrovascular, respiratory, hepatic, renal, GI, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the IP; or may interfere with the interpretation of data

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: Placebo (BW >=50 kg) | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: Placebo (BW <50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: Placebo (BW 40 to 60 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
Started | 3 | 6 | 2 | 7 | 3 | 7
Received At Least One Dose of Study Drug | 2 | 6 | 2 | 7 | 3 | 7
Completed | 2 | 5 | 2 | 6 | 3 | 6
Not Completed | 1 | 1 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Cohort 1: Placebo (BW >=50 kg): Participants in this cohort had a screening body weight of at least 50 kg received placebo administered SC QW during Weeks 1 to 8.
- Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg): Participants in this cohort had a screening body weight of at least 50 kg received 2.5 mg tirzepatide administered SC QW during Weeks 1 to 4 followed by 5 mg tirzepatide during Weeks 5 to 8.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo (BW >=50 kg) | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: Placebo (BW <50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: Placebo (BW 40 to 60 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg) | Total
Number analyzed (Participants) | 2 | 6 | 2 | 7 | 3 | 7 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 6 | 2 | 7 | 3 | 7 | 27
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 5 | 2 | 4 | 17
  Male | 1 | 3 | 0 | 2 | 1 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 0 | 2 | 5
  Not Hispanic or Latino | 2 | 5 | 2 | 5 | 3 | 5 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 2 | 2 | 1 | 4 | 14
  White | 1 | 2 | 0 | 5 | 2 | 3 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 2 | 7 | 3 | 7 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs)
Description: Percentage of participants with TEAEs and SAEs were reported here. A summary of TEAEs, SAEs and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events section of this record.
Time Frame: Baseline through Week 14
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: Placebo (BW >=50 kg) | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: Placebo (BW <50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: Placebo (BW 40 to 60 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
Number analyzed (Participants) | 2 | 6 | 2 | 7 | 3 | 7
Percentage of participants
  TEAE | 0.0 | 83.3 | 0.0 | 85.7 | 33.3 | 100.0
  SAE | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to the End of the Dosing Interval (AUC0-tau) of Tirzepatide
Description: PK: AUC0-tau of tirzepatide was reported.
Time Frame: Predose on weeks 3, 6, 8; 12 and 24 hours post first dose; Within 24 to 96 hours post-dose at week 4; Within 120 to 168 hours post-dose at week 6.
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanogram *hour per milliliter (ng*h/mL)
Arm/Group | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
Number analyzed (Participants) | 6 | 7 | 7
nanogram *hour per milliliter (ng*h/mL) | 105000 (33100) | 80800 (9580) | 156000 (22500)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of Tirzepatide
Description: PK: Cmax of tirzepatide
Time Frame: as for outcome 2
Population: All participants who received at least one dose of tirzepatide and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
Number analyzed (Participants) | 6 | 7 | 7
nanograms per milliliter (ng/mL) | 884 (243) | 674 (63.8) | 1280 (194)

ADVERSE EVENTS:
Time Frame: Baseline Up To 14 Weeks
Description: All participants who received at least one dose of study drug. Per protocol, Adverse Event analysis was planned as per treatment regimen received.
Groups:
- Cohort 1: Placebo (BW >=50 kg): Participants in this cohort had a screening body weight of at least 50 kilograms (kg) received placebo administered subcutaneously (SC) once weekly (QW) in Weeks 1 to 8.
- Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg): Participants in this cohort had a screening body weight of at least 50 kg received 2.5 milligrams (mg) tirzepatide administered SC QW in Weeks 1 to 4 followed by 5 mg tirzepatide in Weeks 5 to 8.
- Cohort 2: Placebo (BW <50 kg): Participants in this cohort had a screening body weight less than 50 kg received placebo administered SC QW in Weeks 1 to 8.
- Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg): Participants in this cohort had a screening body weight less than 50 kg received 1.25 mg tirzepatide administered SC QW in Weeks 1 to 4 followed by 2.5 mg tirzepatide in Weeks 5 to 8.
- Cohort 3: Placebo (BW 40 to 60 kg): Participants in this cohort had a screening body weight between 40 to 60 kg, inclusive, received placebo administered SC QW in Weeks 1 to 8.
- Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg): Participants in this cohort had a screening body weight between 40 to 60 kg, inclusive, received 2.5 mg tirzepatide administered SC QW in Weeks 1 to 4 followed by 5 mg tirzepatide in Weeks 5 to 8.
Arm/Group | Cohort 1: Placebo (BW >=50 kg) | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) | Cohort 2: Placebo (BW <50 kg) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) | Cohort 3: Placebo (BW 40 to 60 kg) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/7 | 0/3 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/2 | 0/7 | 0/3 | 0/7
Other Adverse Events (participants affected / at risk) | 0/2 | 5/6 | 0/2 | 6/7 | 1/3 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (BW >=50 kg) (N=2) | Cohort 1: 2.5-5 mg Tirzepatide (BW >=50 kg) (N=6) | Cohort 2: Placebo (BW <50 kg) (N=2) | Cohort 2: 1.25-2.5 mg Tirzepatide (BW <50 kg) (N=7) | Cohort 3: Placebo (BW 40 to 60 kg) (N=3) | Cohort 3: 2.5-5 mg Tirzepatide (BW 40 to 60 kg) (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (5) | 4 (9)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (11)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT05696847/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05696847/SAP_001.pdf